CLINICAL TRIAL: NCT06126068
Title: Comparison of Loading Dose Magnesium Sulphate With Prichard Regimen in the Management of Severe Preeclampsia and Eclampsia in a Resource Poor Setting, Southeast Nigeria.
Brief Title: Comparison of Loading Dose Magnesium Sulphate With Prichard Regimen in the Management of Severe Preeclampsia and Eclampsia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Nwali Matthew Igwe, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSPL2023CT
Record Dates: First submitted 2023-11-03; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Severe Pre-eclampsia; Eclampsia
Keywords: Pre-eclampsia; Eclampsia; magnesium sulphate
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Intervention Model Description: Prevention of Eclampsia in severe pre-eclampsia and further fits in Eclampsia.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first arm - Loading dose of magnesium sulfate (Active Comparator): This arm received Loading dose of magnesium sulfate only. those that developed complication in each arm were managed according to departmental protocol.
  Interventions: Drug: Use of magnesium sulfate to prevent and stop fits in pre-eclampsia and Eclampsia
- 2. Pritchard regimen (Active Comparator): This arm received the full dose of magnesium sulfate regimen by Pritchard. those that developed complication in each arm were managed according to departmental protocol also.
  Interventions: Drug: Use of magnesium sulfate to prevent and stop fits in pre-eclampsia and Eclampsia

INTERVENTIONS:
Drug: Use of magnesium sulfate to prevent and stop fits in pre-eclampsia and Eclampsia — Loading dose magnesium sulfate versus the Pritchard regimen

SUMMARY:
Preeclampsia/eclampsia is part of a spectrum of multi-systemic pregnancy disorder that contributes substantially to maternal and perinatal morbidity and mortality, especially in low resource setting. This study was done in Abakaliki, Ebonyi State, Southeast Nigeria.

To compare the efficacy of loading dose of magnesium sulphate with that of the Pritchard regimen in the prevention of eclampsia in severe preeclampsia and recurrent fits in eclampsia in a low resource setting.

A prospective, single blinded randomized controlled study of loading dose versus Pritchard regimens of MgSO4 at the Teaching Hospital Abakaliki. One hundred and twenty patients were recruited 60 to each arm using computer-generated numbers. Sociodemographic characteristics, efficacy and adverse effects of the drug on the mother and baby were noted.

DETAILED DESCRIPTION:
Background: Preeclampsia/eclampsia is part of a spectrum of multi-systemic pregnancy disorder that contributes substantially to maternal and perinatal morbidity and mortality, especially in low resource setting. This study was done in Abakaliki, Ebonyi State, Southeast Nigeria.

Objectives: To compare the efficacy of loading dose of magnesium sulphate with that of the Pritchard regimen in the prevention of eclampsia in patients with severe preeclampsia and recurrent fits in eclampsia in a low resource setting like ours.

Methods: This was a prospective, single blinded randomized controlled study of loading dose versus Pritchard regimens of MgSO4 at Alex Ekwueme Federal University Teaching Hospital Abakaliki. One hundred and twenty patients were recruited 60 to each arm using computer-generated numbers. Social demographic characteristics, efficacy and adverse effects of the drug on the mother and baby were noted. Data were collated, tabulated and analyzed using the statistical package for social sciences (SPSS) software (version 22, Chicago II, USA)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with severe preeclampsia
* Pregnant women with eclampsia
* Signing of informed consented to participate in the study.

Exclusion Criteria:

* Refusal of consent,
* Gestational age < 28 weeks
* Received magnesium sulphate prior to presentation
* mild preeclampsia
* chronic hypertension in pregnancy
* Medical or Obstetrical complication of pregnancy.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of convulsions | During the intervention
  percentage of fits in severe pre-eclampsia and recurrence of fits in eclampsia

SECONDARY OUTCOMES:
Drug toxicity | During the intervention
  number of neonatal asphyxia, respiratory depression, loss of tendon reflex and cardiac arrest.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Teaching Hospital, Abakaliki, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No